CLINICAL TRIAL: NCT05504421
Title: The Effect of Cooperative Learning Based Simulation Practice on Nursing Students' Knowledge, Skills and Attitudes Towards Sustainability in Care
Brief Title: The Effect of Cooperative Learning Based Simulation Practice on Sustainability in Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Nagihan Ilaslan, Principal Investigator, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DuzceU-Ilaslan-001
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Nursing Education Research; Nursing Students
Keywords: Nursing students; Simulation; Cooperative learning; Sustainability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Students will receive theoretical training on sustainability in nursing, given by the narrative technique, and then students will work individually on the subject and share their weekly individual study time with the researcher. When individual work is completed, a simulation application will be performed with the scenario.
  Interventions: Other: Sustainability education in nursing to be given with two different teaching methods
- Experimental group (Experimental): Students will receive theoretical training on sustainability in nursing, given by the narrative technique, and then analyze the some structured cases in groups structured in line with the cooperative learning process. When the case analysis is finished, a simulation application will be performed with the scenario.
  Interventions: Other: Sustainability education in nursing to be given with two different teaching methods

INTERVENTIONS:
Other: Sustainability education in nursing to be given with two different teaching methods — Sustainability education in nursing to be given with two different teaching methods (cooperative learning versus traditional learning) and the effects of two different teaching methods on the sustainability knowledge, attitude and skill acquisition of nursing students will be compared.

SUMMARY:
Nurses, who are an individual interacting with their environment, a professional member of the nursing profession providing uninterrupted care to people, and a part of society, are in a very important position in terms of reshaping the interaction of people with environment.

For this, they should be supported to gain cognitive and affective competence on issues such as holistic health understanding and relationship between sustainability and nursing care during nursing education.

The planned study aims to evaluate the effect of simulation practice based on cooperative learning on developing knowledge, skills and attitudes in nursing students about sustainability in nursing care.

The universe of the study, which was planned as a randomized controlled study in an experimental design, will consist of 3rd year nursing students at Düzce University, Department of Nursing.

Data will be collected using the Descriptive Characteristics Form, Nursing Sustainability Information Form, the Debriefing Session Form, Sustainability Attitudes in Nursing Survey (SANS-2), and Ecocentric, Anthropocentric and Antipathic Attitude Toward Environment Scale.

DETAILED DESCRIPTION:
Introduction: Human health should be considered together with the living and non-living environment in which it interacts in the ecosystem. Nurses, who are an individual interacting with their environment, a professional member of the nursing profession providing uninterrupted care to people, and a part of society, are in a very important position in terms of reshaping the interaction of people with environment. At the same time, the nursing ethics codes updated by ICN in 2021 reveal the responsibilities of nurses in the protection and development of global health as a necessity.

However, in order to be able to fulfill their roles and responsibilities, they must first be aware of the necessity of being sustainable in the interaction beings with their environment and understand the impact of their care practices on environmental sustainability. For this, they should be supported to gain cognitive and affective competence on issues such as holistic health understanding, sustainability, the relationship between sustainability and nursing care during nursing education.

Aim:The planned study aims to evaluate the effect of simulation practice based on cooperative learning on developing knowledge, skills and attitudes in nursing students about sustainability in nursing care.

Theoretical framework: In line with the purpose determined within the scope of the study, the simulation practice will be structured in line with the cooperative learning process. Cooperative learning, which is based on the Social Constructivism Theory, founded by John Dewey and Vygotsky, attaches importance to social and individual differences in learning and sees learning as a product of the social interaction process.

Method: The universe of the study, which was planned as a randomized controlled study in an experimental design, will consist of 212 nursing students studying at the 3rd grade level at Düzce University, Department of Nursing in the Fall Semester of the 2022-2023 Academic Year. The number of students to be included in the study sample was calculated as 64 students based on power analysis, and 70 students will form the study sample, taking into account the losses that may occur during the study. Simple random sampling method will be used to determine the students to be included in the study.

Data will be collected using the Descriptive Characteristics Form (10 questions such as age, gender), Nursing Sustainability Information Form (5 open-ended questions), the Debriefing Session Form (the form shaped by the PEARLS depriefing method will be used after simulation), the Sustainability Attitudes in Nursing Survey (SANS-2) (7-point Likert scale containing 9 items), and Ecocentric, Anthropocentric and Antipathic Attitude Toward Environment Scale (7-point Likert scale containing 26 items). The permission to use scales has been obtained from authors via e-mail.

The first measurement will be made in both the experimental and control groups using data collection forms (Descriptive Characteristics Form, Nursing Sustainability Information Form, Sustainability Attitudes in Nursing Survey (SANS-2) and Ecocentric, Anthropocentric and Antipathic Attitude Toward Environment Scale). Then, both groups will be informed in the same session with a 90-minute lecture on sustainability in nursing prepared in line with the NurSus Project resources (http://nursus.eu/home). After this stage, the experimental group students will experience 4-weeks cooperative learning process (will be used the Group Research Technique) that aims to analysis cases related to sustainability in nursing (cases were shaped in line with the resources in the NurSus Project). The control group will work individually on the subject and share their weekly individual study time with the researcher. After the case analysis process, simulation practice will be carried out in line with the a scenario with both groups. Simulation practice aims to develop the students' ability to transfer their sustainability knowledge and attitudes on nursing skills. And the second measurement will be carried out immediately after the simulation practice (Nursing Sustainability Information Form, Sustainability Attitudes in Nursing Survey (SANS-2), Ecocentric, Anthropocentric and Antipathic Attitude Toward Environment Scale and Debriefing Session Form).

In the analysis of the data, within and between group comparisons will be conducted. So, the effect of two different teaching methods (cooperative learning and traditional learning) on gaining nursing students sustainability knowledge, attitudes and skills will be compared.

ELIGIBILITY:
Inclusion Criteria:

* 3rd year nursing student
* Volunteering to participate in the study

Exclusion Criteria:

-Not wanting to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Sustainability Attitudes in Nursing Survey (SANS-2) | a day before the training
  Students will mark the level of participation for each item (total 9 item)in the 7-point likert scale.
Sustainability Attitudes in Nursing Survey (SANS-2) | one hour after the simulation application
  Students will mark the level of participation for each item (total 9 item) in the 7-point likert scale.
Sustainability Attitudes in Nursing Survey (SANS-2) | one year after the training
  Students will mark the level of participation for each item (total 9 item)in the 7-point likert

SECONDARY OUTCOMES:
Descriptive Characteristics Form | a day before the training
  Students will answer questions about descriptive characteristics such as age and gender.
Nursing Sustainability Information Form | a day before the training
  Students will answer open-ended questions about sustainability in nursing care.
Nursing Sustainability Information Form | one hour after the simulation application
  Students will answer open-ended questions about sustainability in nursing care.
Ecocentric, Anthropocentric and Antipathic Attitude Toward Environment Scale | a day before the training
  Students will mark the level of participation for each item (total 26 item) in the 7-point likert scale.
Ecocentric, Anthropocentric and Antipathic Attitude Toward Environment Scale | one hour after the simulation application
  Students will mark the level of participation for each item (total 26 item) in the 7-point likert scale.
Debriefing Session Form | one hour after the simulation application
  After the simulation application, a debriefing session will be conducted with the students in line with open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Nagihan İlaslan, MSc, Principal Investigator — Duzce University; Nuray Şahin Orak, PhD, Principal Investigator — Istanbul Nisantasi University
Locations (1):
- Duzce University, Düzce, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilaslan N, Sahin Orak N. Sustainable healthcare education using cooperative simulation in developing nursing students' knowledge, attitude and skills: A randomized controlled study. Nurse Educ Today. 2025 Aug;151:106706. doi: 10.1016/j.nedt.2025.106706. Epub 2025 Mar 20. PMID 40139038